CLINICAL TRIAL: NCT07256496
Title: Enhanced Dialectical Behavior Therapy for Adolescents: Impacts of Individualized Skills Coaching on Constructs of Suicidality
Brief Title: Enhanced Dialectical Behavior Therapy for Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Compass Behavioral Health (Other)
Responsible Party: Principal Investigator, Megan Plakos Szabo, Associate Director of Research, Compass Behavioral Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00078098
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Suicidality
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enhanced DBT-A Group (Experimental): Participants engaged in Enhanced DBT-A services, including individual therapy, group skills training, phone coaching, and ISCS. Participants completed assessment batteries at intake, 6 months, and 1 year, and the outcome measures assessed participants' severity and intensity of suicidal ideation (SI), reasons for living, and depressive symptoms.
  Interventions: Behavioral: Enhanced DBT-A

INTERVENTIONS:
Behavioral: Enhanced DBT-A — Participants engaged in Enhanced DBT-A services, including individual therapy, group skills training, phone coaching, and ISCS. Participants completed assessment batteries at intake, 6 months, and 1 year, and the outcome measures assessed participants' severity and intensity of suicidal ideation (SI), reasons for living, and depressive symptoms.

SUMMARY:
Suicide is a leading cause of death and significant concerns for adolescents and young adults. Dialectical Behavior Therapy for Adolescents (DBT-A) is an evidence-based intervention that effectively reduces life-threatening behaviors. Limited research examines the impact of adding individualized skills coaching sessions (ISCS) to the DBT-A model, a novel intervention referred to in this paper as "Enhanced DBT-A". This study evaluates the effectiveness of Enhanced DBT-A in reducing suicidality over 1 year of treatment in an outpatient and intensive outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* appropriateness for Stage 1 DBT, completion of all assessments within the designated timeframe, a non-zero score on the Columbia-Suicide Severity Rating Scale (C-SSRS) at intake, and participation in at least one ISCS between intake and 1 year from the first individual therapy session.

Exclusion Criteria:

* presenting with active psychosis, a primary diagnosis of substance use, who did not consent to data collection, or who had a zero score on the C-SSRS at intake

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2014-10-17 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Reasons for Living Inventory for Adolescents (RFL-A) | 1 year
  The Reasons for Living Inventory for Adolescents (RFL-A; Osman et al, 1998) is a 32-item self-report questionnaire that assesses adaptive reasons that may prevent an adolescent from engaging in life-threatening behavior.
PHQ-9 | 1 year
  The current study administered the PHQ-9 to participants 18 years and older. The PHQ-9 (Kroenke et al, 2001) is a widely-used and psychometrically-robust self-report measure used to assess the prevalence of depressive symptoms in adults during a two-week period.
Columbia-Suicide Severity Rating Scale - Self Report Screener - Recent (C-SSRS). | 1 year
  To capture the severity and intensity of participants' SI and their corresponding suicide risk, we used items from the Columbia-Suicide Severity Rating Scale - Screen Version - Recent (C-SSRS; Posner et al, 2011).

CONTACTS AND LOCATIONS:
Locations (1):
- Compass Behavioral Health, Tustin, California, United States

IPD SHARING:
Plan to Share IPD: No